CLINICAL TRIAL: NCT05244226
Title: Pediatric Pain Optimization After Tonsillectomy: A Randomized Double Blind Methadone Pilot Study
Brief Title: Pediatric Pain Optimization After Tonsillectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00109911
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea; Tonsillitis; Pain, Procedural
MeSH Terms: conditions — Sleep Apnea, Obstructive; Tonsillitis; Pain, Procedural | interventions — Fentanyl; Hydromorphone; Methadone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Short acting opioids: Fentanyl, Hydromorphone (Active Comparator)
  Interventions: Drug: Fentanyl/Hydromorphone
- Long Acting Opioid: Methadone (Active Comparator)
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Fentanyl/Hydromorphone — Per routine care
  Arms: Short acting opioids: Fentanyl, Hydromorphone
Drug: Methadone — Initial dosing 0.1mg/kg, potential to escalate to 0.15mg/kg following interim analysis
  Arms: Long Acting Opioid: Methadone

SUMMARY:
The purpose of this study is to compare the use of short acting opioids (fentanyl/hydromorphone) with long acting opioids (methadone) for pain control following tonsillectomy surgery.

DETAILED DESCRIPTION:
This is a single center, randomized, double blind, parallel-group dose escalation investigation which will compare post operative pain control indices for patients receiving short acting versus long acting opioids as intraoperative analgesics. Surgical and anesthesia care, except for intraoperative opioid management, are not altered for study purposes. Subjects are randomized 2:1 to either long-duration (methadone) or short-duration opioid (fentanyl, hydromorphone) through the perioperative period. Exploratory data will be collected for up to 30 days post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3 to 17 years old
* Presenting for elective tonsillectomy +/- adenoidectomy
* Provide informed consent / assent (as appropriate)

Exclusion Criteria:

* History of liver or kidney disease
* Females with positive pregnancy test
* Severe sleep apnea (Sleep study with Apnea Hypopnea Index (AHI) > 10)
* Consistent daily opioid use for chronic pain ( >3 months)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Einhorn, MD, Principal Investigator — Duke University
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Einhorn LM, Hoang J, La JO, Kharasch ED. Single-dose Intraoperative Methadone for Pain Management in Pediatric Tonsillectomy: A Randomized Double-blind Clinical Trial. Anesthesiology. 2024 Sep 1;141(3):463-474. doi: 10.1097/ALN.0000000000005031. PMID 38669011

RESULTS

PARTICIPANT FLOW:
Groups:
- Long Acting Opioid: Methadone 0.1mg/kg: Low dose methadone: 0.1mg/kg
- Long Acting Opioid: Methadone 0.15mg/kg: High dose methadone: 0.15 mg/kg
Period: Overall Study
Arm/Group | Short Acting Opioids: Fentanyl, Hydromorphone | Long Acting Opioid: Methadone 0.1mg/kg | Long Acting Opioid: Methadone 0.15mg/kg
Started | 21 | 22 | 23
Completed | 20 | 20 | 20
Not Completed | 1 | 2 | 3
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Long Acting Opioid: Methadone 0.15mg/kg: High dose methadone: 0.15mg/kg
- Total: Total of all reporting groups
Arm/Group | Short Acting Opioids: Fentanyl, Hydromorphone | Long Acting Opioid: Methadone 0.1mg/kg | Long Acting Opioid: Methadone 0.15mg/kg | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 4.0 [3.0 to 6.3] | 4.5 [4.0 to 6.3] | 4.5 [3.8 to 7.0] | 4.3 [3.6 to 6.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 9 | 30
  Male | 13 | 6 | 11 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 3 | 8
  Not Hispanic or Latino | 18 | 17 | 17 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 6 | 10
  White | 11 | 18 | 12 | 41
  More than one race | 4 | 1 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Total Amount of Opioid Medications Administered
Description: Postoperative opioid medication expressed in oral morphine equivalents (OME) per kilogram
Time Frame: Up to 7 days post surgery
Measure: Median (Inter-Quartile Range); unit: morphine mg equivalents/kg
Groups:
- Long Acting Opioid: Methadone (0.1mg/kg): Low dose methadone: 0.1mg/kg
- Long Acting Opioid: Methadone (0.15mg/kg): High dose methadone: 0.15 mg/kg
Arm/Group | Short Acting Opioids: Fentanyl, Hydromorphone | Long Acting Opioid: Methadone (0.1mg/kg) | Long Acting Opioid: Methadone (0.15mg/kg)
Number analyzed (Participants) | 20 | 20 | 20
morphine mg equivalents/kg | 1.5 [1.2 to 2.1] | 0.9 [0.1 to 1.4] | 0.5 [0 to 1.4]
Statistical Analysis 1: Comparison: Short Acting Opioids: Fentanyl, Hydromorphone vs Long Acting Opioid: Methadone (0.1mg/kg); Test type: Superiority; p = 0.045, Kruskal-Wallis; Dunn's Kruskal Wallis with Bonferroni correction
Statistical Analysis 2: Comparison: Short Acting Opioids: Fentanyl, Hydromorphone vs Long Acting Opioid: Methadone (0.15mg/kg); Test type: Superiority; p = 0.023, Kruskal-Wallis; Dunn's Kruskal Wallis with Bonferroni correction

2. Secondary Outcome: Percentage of Scores on the Parent Post Operative Pain Measure (PPPM) That Indicate Clinically Significant Pain
Description: The PPPM has 15 yes/no questions which results in a score from 0-15, where a higher score indicates greater pain. A score of at least 6 out of 15 signifies clinically significant pain. The percentage of scores > or = 6 is shown below.
Time Frame: Up to 7 days post surgery
Population: Participants who were less than 13 years of age. Each participant reported 7 scores.
Measure: Number; unit: percentage of PPPM scores
Units Other Than Participants: PPPM scores
Groups:
- Long Acting Opioid: Methadone 0.1mg/kg: Low dose methadone 0.1mg/kg
- Long Acting Opioid: Methadone 0.15mg/kg: High dose methadone 0.15mg/kg
Arm/Group | Short Acting Opioids: Fentanyl, Hydromorphone | Long Acting Opioid: Methadone 0.1mg/kg | Long Acting Opioid: Methadone 0.15mg/kg
Number analyzed (Participants) | 19 | 18 | 18
Number analyzed (PPPM scores) | 133 | 126 | 126
percentage of PPPM scores | 57 | 61 | 63

3. Secondary Outcome: NIH PROMIS (Patient-Reported Outcomes Measurement Information System) Parent Proxy Report Scale
Description: Patient caregiver (as proxy) pain scores over past 7 days. Scale of 1 to 6, where 1=had no pain and 6=almost always had pain.
Time Frame: Up to 7 days post surgery
Population: Participants who were less than 13 years of age.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Short Acting Opioids: Fentanyl, Hydromorphone | Long Acting Opioid: Methadone 0.1mg/kg | Long Acting Opioid: Methadone 0.15mg/kg
Number analyzed (Participants) | 19 | 18 | 18
score on a scale | 2.4 (1.5) | 2.2 (1.2) | 2.3 (1.1)

4. Secondary Outcome: Evaluation of Participant's Pain as Measured by Numeric Pain Rating Scale
Description: Numeric Pain Rating Scale has a range of 0 to 10, where 0=no pain and 10=worst possible pain.
Time Frame: Up to 7 days post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Short Acting Opioids: Fentanyl, Hydromorphone | Long Acting Opioid: Methadone (0.1mg/kg) | Long Acting Opioid: Methadone (0.15mg/kg)
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 4.0 (2.5) | 3.7 (1.9) | 3.8 (2.3)

5. Secondary Outcome: Doses of Prescription Opioid Used Following Hospital Discharge
Description: Number of doses of prescription medication used.
Time Frame: Up to 7 days post surgery
Measure: Median (Inter-Quartile Range); unit: doses
Arm/Group | Short Acting Opioids: Fentanyl, Hydromorphone | Long Acting Opioid: Methadone (0.1mg/kg) | Long Acting Opioid: Methadone (0.15mg/kg)
Number analyzed (Participants) | 20 | 20 | 20
doses | 4 [3 to 9] | 2 [0 to 4] | 3 [0 to 5]
Statistical Analysis 1: Comparison: Short Acting Opioids: Fentanyl, Hydromorphone vs Long Acting Opioid: Methadone (0.1mg/kg); Test type: Superiority; p = 0.144, Kruskal-Wallis
Statistical Analysis 2: Comparison: Short Acting Opioids: Fentanyl, Hydromorphone vs Long Acting Opioid: Methadone (0.15mg/kg); Test type: Superiority; p = 0.322, Kruskal-Wallis

6. Secondary Outcome: Opioid Administration in the PACU (Post-anesthesia Care Unit)
Description: Opioid medication use in the recovery room expressed in oral morphine equivalents (OME) per kilogram.
Time Frame: Up to 6 hours post surgery
Measure: Median (Inter-Quartile Range); unit: morphine mg equivalents/kg
Arm/Group | Short Acting Opioids: Fentanyl, Hydromorphone | Long Acting Opioid: Methadone (0.1mg/kg) | Long Acting Opioid: Methadone (0.15mg/kg)
Number analyzed (Participants) | 20 | 20 | 20
morphine mg equivalents/kg | 0.15 [0.10 to 0.30] | 0.04 [0 to 0.1] | 0 [0 to 0.1]
Statistical Analysis 1: Comparison: Short Acting Opioids: Fentanyl, Hydromorphone vs Long Acting Opioid: Methadone (0.1mg/kg); Test type: Superiority; p = 0.061, Kruskal-Wallis; Dunn's Kruskal Wallis with Bonferroni correction
Statistical Analysis 2: Comparison: Short Acting Opioids: Fentanyl, Hydromorphone vs Long Acting Opioid: Methadone (0.15mg/kg); Test type: Superiority; p = 0.021, Kruskal-Wallis; Dunn's Kruskal Wallis with Bonferroni correction

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Short Acting Opioids: Fentanyl, Hydromorphone | Long Acting Opioid: Methadone (0.1mg/kg) | Long Acting Opioid: Methadone (0.15mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Short Acting Opioids: Fentanyl, Hydromorphone (N=21) | Long Acting Opioid: Methadone (0.1mg/kg) (N=22) | Long Acting Opioid: Methadone (0.15mg/kg) (N=23)
Altered mental status (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/26/NCT05244226/Prot_SAP_000.pdf